CLINICAL TRIAL: NCT02576119
Title: A Randomized, Double-Blind, Double-Dummy, Positive-Controlled, Crossover Study to Determine Electrocardiographic Effects of BMS-955176 in Healthy Subjects
Brief Title: A Study to Determine the Effect of Multiple Doses of BMS-955176 on the Electrocardiograph of Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated early due to neuropsychiatric serious adverse events reported by 2 participants.
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 206220; AI468-044 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — BMS-955176; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Sentinal Cohorts (Experimental): Study is in 2 sequential cohorts (BMS-955176 or placebo) each to evaluate the safety, tolerability, and PK following multiple-dose administration of BMS-955176.
  Interventions: Drug: BMS-955176, Placebo (Part 1)
- Part 2: Main QTc Study (Experimental): 3 period nested crossover study.
  Interventions: Drug: BMS-955176, Moxifloxacin, Placebo (Part 2)

INTERVENTIONS:
Drug: BMS-955176, Placebo (Part 1) — The BMS-955176 dose in sentinel Cohort 1 will be 240 mg orally. The BMS-955176 dose in sentinel Cohort 2 will be determined based on the results of data from sentinel Cohort 1.
  Arms: Part 1: Sentinal Cohorts
Drug: BMS-955176, Moxifloxacin, Placebo (Part 2) — Subjects will be randomized to 1 of 12 sequences. Each sequence includes combination of different regimens (combination of BMS-955176, placebo and Moxifloxacin).
  Arms: Part 2: Main QTc Study

SUMMARY:
The purpose of the study is to determine the effect of multiple doses of BMS-955176 on the QT interval corrected with Fridericia's method (QTcF) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent
2. Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination findings, 12-lead ECG measurements, physical measurements, and clinical laboratory test results
3. Body mass index (BMI) of 18.0 kg/m2 to 32.0 kg/m2, inclusive, at screening and Day 1. BMI = weight (kg)/[height(m)]2
4. Women must have a negative serum pregnancy test, must not be breastfeeding, and women of child bearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with BMS-955176 in addition to a post-treatment completion period
5. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with BMS-955176 in addition to a post-treatment completion period

Exclusion Criteria:

1. Any significant acute or chronic medical illness
2. Any GI disease or surgery that can affect absorption of the study drug
3. A personal history of clinically relevant cardiac disease, long QT syndrome, symptomatic or asymptomatic arrhythmias, presyncope or syncopal episodes, or additional risk factors for torsades de pointes (eg, heart failure)
4. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population
5. History of allergy to moxifloxacin, HIV maturation inhibitors, or related compounds

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 315 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2016-02-26 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Part 1: Reported adverse events | Selected time points up to 24 hours postdose
Part 1: Vital sign measurements | Selected time points up to 24 hours postdose
Part 1: Physical examinations | Selected time points up to 24 hours postdose
Part 1: Safety 12-lead ECGs | Selected time points up to 24 hours postdose
Part 2: ΔΔQTcF, the subject specific time-matched difference between the ΔQTcF (QT interval corrected with Fridericia's method) after administration of BMS-955176 and the ΔQTcF after administration of placebo | Days 1 to 28

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States